CLINICAL TRIAL: NCT04853901
Title: Remdesivir Efficacy In Management Of COVID-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hany Dabbous, Professor of Tropical Medicine Faculty of Medicine Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU P56a/ 2020
Record Dates: First submitted 2021-03-01; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; Hydroxychloroquine; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remdesivir (Experimental): Remdesivir loading dose of 200 mg intravenously followed by 100 mg/day intravenously for 5 to 10days + Methylprednisolone 1-2mg/kg for 5-7 days
  Interventions: Drug: Remdesivir
- Standard of care therapy (Active Comparator): Hydroxycoloroquine 400mg twice on day 1 then 200mg tab twice 2-10 days + Methylprednisolone 1-2mg/kg for 5-7 days
  Interventions: Drug: Standard of care_1; Drug: Standard of care_2

INTERVENTIONS:
Drug: Remdesivir — Remdesivir loading dose of 200 mg intravenously followed by 100 mg/day intravenously for 5 to 10days
  Other Names: Veklury
  Arms: Remdesivir
Drug: Standard of care_1 — Hydroxycoloroquine 400mg twice on day 1 then 200mg tab twice 2-10 days
  Other Names: Plaquenil
  Arms: Standard of care therapy
Drug: Standard of care_2 — Methylprednisolone 1-2mg/kg for 5-7 days
  Other Names: Steroid
  Arms: Standard of care therapy

SUMMARY:
The study is open label randomized interventional phase 3 clinical trial. Patients with confirmed Covid-19 cases who was hospitalized in Two university isolation hospitals (Ain Shams University and Assiut University ) assigned hospitals for isolation.

DETAILED DESCRIPTION:
The study is open label randomized interventional phase 3 clinical trial. Patients with confirmed Covid-19 cases who was hospitalized in Two university isolation hospitals (Ain Shams University and Assiut University ) assigned hospitals for isolation.

The included patients receive. Intervention group: Remdesivir loading dose of 200 mg intravenously followed by 100 mg/day intravenously for 5 to 10days + Methylprednisolone 1-2mg/kg for 5-7 days Control group: standard of care without Remdesivir

ELIGIBILITY:
Inclusion Criteria:

Adult 18 -80 years old Must have laboratory confirmed COVID-19(A patient with laboratory confirmation (Positive RT-PCR) of COVID-19 infection, irrespective of clinical signs and symptoms according to Ain Shams University Hospitals Consensus Statement on Management of Adult COVID-19 Patients.

Must have severe or immediately life-threatening COVID-19,

* Severe disease is defined as:

  * Dyspnea,
  * Respiratory frequency ≥ 30/min,
  * Blood oxygen saturation ≤ 93%,
  * Partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or lung infiltrates > 50% within 24 to 48 hours
* Life-threatening disease is defined as:

  * respiratory failure,
  * septic shock, and/or
  * multiple organ dysfunction or failure
* Must provide informed consent by patient or his/her legal guardian or Professional Legal Representative

Exclusion Criteria:

* Mild to moderately affected COVID 19 confirmed patients.
* pregnancy, lactation.
* known hepatic failure.
* Patient who is not likely to comply to study procedures.
* Creatine clearance <30 ml/min.
* Elevated transaminases > 5 fold ULN.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of viral clearance | 14 days
  Achievement of two successive negative COVID-19 PCR analysis tests 72 hours apart

CONTACTS AND LOCATIONS:
Overall Officials: Hany E Dabbous, M.D, Principal Investigator — Faculty of Medicine Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No